CLINICAL TRIAL: NCT02535312
Title: Phase I Study of TRC102 in Combination With Cisplatin and Pemetrexed in Patients With Advanced Solid Tumors / Phase II Study of TRC102 With Pemetrexed in Patients Refractory to Pemetrexed and Cisplatin or Carboplatin
Brief Title: Methoxyamine, Cisplatin, and Pemetrexed Disodium in Treating Patients With Advanced Solid Tumors or Mesothelioma That Cannot Be Removed by Surgery or Mesothelioma That Is Refractory to Pemetrexed Disodium and Cisplatin or Carboplatin
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00127; NCI-2015-00127 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-76; 9837 (Other: City of Hope Comprehensive Cancer Center LAO); 9837 (Other: CTEP); UM1CA186689 (NIH); UM1CA186705 (NIH); UM1CA186717 (NIH); ZIABC011078 (NIH)
Record Dates: First submitted 2015-08-27; First posted 2015-08-28 (Estimated); Results first posted 2024-04-25 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Solid Neoplasm; Advanced Peritoneal Malignant Mesothelioma; Advanced Pleural Malignant Mesothelioma; Recurrent Peritoneal Malignant Mesothelioma; Recurrent Pleural Malignant Mesothelioma; Refractory Malignant Solid Neoplasm; Unresectable Solid Neoplasm
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; methoxyamine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (methoxyamine, pemetrexed disodium, cisplatin) (Experimental): Patients receive methoxyamine PO QD on days 1-4, pemetrexed disodium IV over 10 minutes, and cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue methoxyamine and pemetrexed disodium beyond cycle 6 if the patient continues to benefit from treatment at the discretion of the treating physician.
  Interventions: Drug: Cisplatin; Drug: Methoxyamine; Drug: Pemetrexed Disodium
- Arm B (methoxyamine, pemetrexed disodium) (Experimental): Patients receive methoxyamine PO QD on days 1-4 and pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue methoxyamine and pemetrexed disodium beyond cycle 6 if the patient continues to benefit from treatment at the discretion of the treating physician.
  Interventions: Drug: Methoxyamine; Drug: Pemetrexed Disodium

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm A (methoxyamine, pemetrexed disodium, cisplatin)
Drug: Methoxyamine — Given PO
  Other Names: TRC102 Base
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; Almita; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt

SUMMARY:
This phase I/II trial studies the side effects and the best dose of methoxyamine when given together with cisplatin and pemetrexed disodium and to see how well it works in treating patients with solid tumors or mesothelioma that have spread to other places in the body and usually cannot be cured or controlled with standard treatment (advanced), or mesothelioma that does not respond to pemetrexed disodium and cisplatin or carboplatin (refractory). Methoxyamine may shrink the tumor and may also help cisplatin and pemetrexed disodium work better by making tumor cells more sensitive to the drugs. Drugs used in chemotherapy, such as cisplatin and pemetrexed disodium, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving methoxyamine together with cisplatin and pemetrexed disodium may be a better treatment for solid tumors or mesothelioma than methoxyamine and pemetrexed disodium.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) for the combination of methoxyamine (TRC102) with pemetrexed (pemetrexed disodium) and cisplatin in patients with advanced solid tumors. (Arm A) II. To describe the toxicities of TRC102 combined with pemetrexed and cisplatin at each dose studied. (Arm A) III. To describe responses to the drug combination at each dose level. (Arm A) IV. To detect activity of the combination of TRC102 and pemetrexed, as evidenced by tumor response in patients with advanced malignant mesothelioma previously treated with pemetrexed and cisplatin. (Arm B)

SECONDARY OBJECTIVES:

I. To describe pharmacokinetic parameters of TRC102 given concurrent with pemetrexed and cisplatin.

II. To evaluate the pharmacodynamic parameters of TRC102 given concurrently with pemetrexed and cisplatin.

III. To explore the feasibility of establishing pleural and peritoneal effluent-derived cell lines and to evaluate the response of cultured pleural and peritoneal mesothelioma cells to cisplatin, pemetrexed, and TRC102.

IV. To document all objective clinical responses to TRC102 in combination with pemetrexed and cisplatin.

OUTLINE: This is a phase I, dose-escalation study of methoxyamine, followed by a phase II study. Patients are assigned to 1 of 2 treatment arms.

ARM A: Patients receive methoxyamine orally (PO) once daily (QD) on days 1-4, pemetrexed disodium intravenously (IV) over 10 minutes, and cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue methoxyamine and pemetrexed disodium beyond cycle 6 if the patient continues to benefit from treatment at the discretion of the treating physician.

ARM B: Patients receive methoxyamine PO QD on days 1-4 and pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue methoxyamine and pemetrexed disodium beyond cycle 6 if the patient continues to benefit from treatment at the discretion of the treating physician.

After completion of study treatment, patients are followed up for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Arm A dose escalation: patients with histologically or cytologically proven advanced solid tumors for which standard treatments are not available, or for whom the current dose level of cisplatin in combination with pemetrexed is appropriate; =< 2 prior cytotoxic chemotherapy regimen
* Arm A dose level 4 (75 mg/m^2 cisplatin): patients with histologically proven chemotherapy-naive advanced unresectable solid tumors for which pemetrexed combined with cisplatin is an indicated regimen
* Arm B (first stage of phase II of TRC102 and pemetrexed): patients with malignant pleural or peritoneal mesothelioma who had progressed while being treated with or had recurred within 6 months of being treated with pemetrexed and cisplatin or carboplatin frontline; intervening treatment is allowed
* Prior pemetrexed is allowed except Arm A dose level 4 (cisplatin 75 mg/m^2)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 -1 (Karnofsky >= 70%)
* Life expectancy of greater than 3 months
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 10.0 g/dl
* Prothrombin time or international normalized ratio (INR) =< 1.5 x upper limit of normal (ULN)
* Total bilirubin < 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN or =< 5 x ULN if metastatic disease involves liver
* Serum creatinine =< 1.5 x ULN or a calculated creatinine clearance >= 60 ml/min/1.73 m^2 (Cockcroft-Gault method) for patients receiving combination of cisplatin and pemetrexed and >= 45 ml/min/1.73 m^2 for patients receiving pemetrexed; 24 hour urine for creatinine clearance is acceptable if the calculated creatinine clearance is insufficient
* For patients enrolled in Arm B (first stage of phase II of TRC102 and pemetrexed) measurable disease is required according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria for patients with solid tumors and modified RECIST criteria as described by Byrne and Novak for patients with malignant pleural mesothelioma; pleural effusion and ascites are not considered measurable disease
* Patients must be able to swallow whole capsules; nasogastric or gastrointestinal (G)-tube administration is not allowed
* The effects of TRC102 on the developing human fetus are unknown; for this reason and because TRC102 as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of the study drugs; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of TRC102, pemetrexed and cisplatin administration; non-childbearing potential is defined as (by other than medical reasons): >= 45 years of age and has not had menses for >= 2 years, amenorrheic for < 2 years without hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation, or post hysterectomy, oophorectomy or tubal ligation; documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by ultrasound; tubal ligation must be confirmed with medical records of the actual procedure otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit though 4 months after the last dose of study drugs
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; patients who have had targeted therapy will be required to wait 2 weeks due to short half-life of the drugs; treatment with bisphosphonates is permitted
* Patients who are receiving any other investigational agents
* Patients with active brain metastases or carcinomatous meningitis are excluded from this clinical trial; patients with treated brain metastases, whose brain metastatic disease has remained stable for greater than or equal to 4 weeks without requiring steroid and anti-seizure medications are eligible to participate
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TRC102 or pemetrexed and cisplatin
* No studies have been performed to assess potential metabolic and transport interactions of TRC102; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product; the case report form must capture the concurrent use of all other drugs, over-the-counter medications, or alternative therapies
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because TRC102 is agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with TRC102, breastfeeding should be discontinued if the mother is treated with TRC102; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with TRC102; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients with known disorders associated with hemolysis
* Patients with thromboembolic disease and on anticoagulation
* Patients with a prior cumulative cisplatin dose > 300 mg/m^2 (pertains to Arm A only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-10-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Koczywas, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (14):
- United States (14):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A, Dose Level 1 - 50mg TRC102, 60mg/m^2 Cisplatin (Phase I): TRC102 50 mg/day PO days 1-4; Pemetrex 500 mg/m^2 IV over 10 min day1; Cisplatin 60 mg/m^2 IV over 30-60 min day1
- Arm A, Dose Level 2 - 75mg TRC102, 60mg/m^2 Cisplatin (Phase I): TRC102 75 mg/day PO days 1-4; Pemetrex 500 mg/m^2 IV over 10 min day1; Cisplatin 60 mg/m^2 IV over 30-60 min day1
- Arm A, Dose Level 3 - 100mg TRC102, 60mg/m^2 Cisplatin (Phase I): TRC102 100 mg/day PO days 1-4; Pemetrex 500 mg/m^2 IV over 10 min day1; Cisplatin 60 mg/m^2 IV over 30-60 min day1
- Arm A, Dose Level 4 - 100mg TRC102, 75mg/m^2 Cisplatin (Phase I): TRC102 100 mg/day PO days 1-4; Pemetrex 500 mg/m^2 IV over 10 min day1; Cisplatin 75 mg/m^2 IV over 30-60 min day1
- Arm B, Dose Level 1 - 50mg TRC102 (Phase II): TRC102 50mg/day PO on days 1-4; Pemetrex 500mg/m^2 IV over 10 min day 1
Period: Overall Study
Arm/Group | Arm A, Dose Level 1 - 50mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 2 - 75mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 3 - 100mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 4 - 100mg TRC102, 75mg/m^2 Cisplatin (Phase I) | Arm B, Dose Level 1 - 50mg TRC102 (Phase II)
Started | 3 | 4 | 3 | 6 | 14
Completed | 3 | 4 | 3 | 6 | 14
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A, Dose Level 3 - 100mg TRC102, 60mg/m^2 Cisplatin (Phase I): TRC102 100 mg/dayPO days 1-4; Pemetrex 500 mg/m^2 IV over 10 min day1; Cisplatin 60 mg/m^2 IV over 30-60 min day1
- Total: Total of all reporting groups
Arm/Group | Arm A, Dose Level 1 - 50mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 2 - 75mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 3 - 100mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 4 - 100mg TRC102, 75mg/m^2 Cisplatin (Phase I) | Arm B, Dose Level 1 - 50mg TRC102 (Phase II) | Total
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 14 | 30
Age, Continuous [Median (Full Range); unit: years] | 69 [60 to 70] | 61.5 [57 to 71] | 66 [65 to 74] | 68.5 [60 to 76] | 74.5 [56 to 85] | 70 [56 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 3 | 3 | 8
  Male | 3 | 3 | 2 | 3 | 11 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 3 | 3 | 4 | 0 | 12
  Hispanic | 1 | 0 | 0 | 1 | 13 | 15
  Unknown | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 3 | 6 | 14 | 30
ECOG performance status [Count of Participants; unit: Participants]
  0=Asymptomatic and fully active | 1 | 3 | 3 | 1 | 3 | 11
  1=Symptomatic; fully ambulatory; restricted in physically strenuous activity | 2 | 1 | 0 | 5 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Dose Limiting Toxicity (DLT) - Phase I
Description: Dose-limiting toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Pre-specified DLT criteria included the following adverse events (AE), judged to be at least possibly related to study therapy: grade 3 or greater non-hematologic toxicity, grade 3 thrombocytopenia with bleeding, any grade 4 thrombocytopenia, grade 4 febrile neutropenia lasting > 7 day, any grade febrile neutropenia, any grade 5 toxicity. Treatment delay of cycle 2 by more than 2 weeks and inability to administer 3 of the 4 doses due to toxicity in the first treatment course were also considered DLTs. Controllable nausea, vomiting and diarrhea, electrolyte toxicities correctable (to baseline or grade 1) with repletion and grade 3 creatinine elevation correctable (to grade 1 or less) with IV hydration were not considered DLT's.
Time Frame: During the first cycle of treatment, up to 21 days
Measure: Count of Participants; unit: Participants
Groups:
- Arm A, Dose Level 3 - 100mg TRC102, 60mg/m^2 Cisplatin (Phase I): TRC102 100/day mg PO days 1-4; Pemetrex 500 mg/m^2 IV over 10 min day1; Cisplatin 60 mg/m^2 IV over 30-60 min day1
- Arm A, Dose Level 4 - 100mg TRC102, 75mg/m^2 Cisplatin (Phase I): TRC102 100/day mg PO days 1-4; Pemetrex 500 mg/m^2 IV over 10 min day1; Cisplatin 75 mg/m^2 IV over 30-60 min day1
Arm/Group | Arm A, Dose Level 1 - 50mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 2 - 75mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 3 - 100mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 4 - 100mg TRC102, 75mg/m^2 Cisplatin (Phase I)
Number analyzed (Participants) | 3 | 4 | 3 | 6
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The maximum tolerated dose of TRC102 in combination with 500mg/m^2 IV of Pemetrex and 60 or 75 mg/m^2 IV of Cisplatin is based on toxicities observed during the first cycle and is defined as the highest dose tested in which fewer than 33% of patients experience an attributable DLT to the study drug, when at least 6 patients are treated at that dose and are evaluable for toxicity. Dose escalations proceeded according to a standard 3+3 design.
Time Frame: 21 days from start of treatment, up to 2 years
Measure: Number; unit: mg/day
Groups:
- Treatment (TRC102, Pemetrexed Disodium, Cisplatin): Patients receive starting dose of TRC102 50 mg/day PO on days 1-4, 500 mg/m^2 pemetrexed disodium IV over 10 minutes, and 60 or 75 mg/m^2 of cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue TRC102 and pemetrexed disodium beyond cycle 6 if the patient continues to benefit from treatment at the discretion of the treating physician.
  Cisplatin: Given IV
  TRC102: Given PO
  Pemetrexed Disodium: Given IV
Arm/Group | Treatment (TRC102, Pemetrexed Disodium, Cisplatin)
Number analyzed (Participants) | 16
mg/day | 100

3. Primary Outcome: Number of Subject With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm; Partial Response (PR), at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; Overall Response (OR) = CR + PR
Time Frame: Up to 8 weeks post-treatment
Measure: Count of Participants; unit: Participants
Groups:
- Arm B, Dose Level 1 - 50mg TRC102 (Phase II): TRC102 50 mg/day PO on days 1-4; Pemetrex 500mg/m^2 IV over 10 min day 1
Arm/Group | Arm A, Dose Level 1 - 50mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 2 - 75mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 3 - 100mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 4 - 100mg TRC102, 75mg/m^2 Cisplatin (Phase I) | Arm B, Dose Level 1 - 50mg TRC102 (Phase II)
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 14
Participants | 0 | 1 | 2 | 0 | 1

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival will be summarized as time from first protocol treatment until progression or death from any cause, using the product-limit Kaplan-Meier estimator. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECISTv1.1), as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From start of treatment to time of progression or death from any cause, whichever occurs first, assessed up to at least 1 year
Population: Pre-specified in the Study Protocol to collect, analyze, and report data for this Outcome Measure by Phase and not by dose-level.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm A (TRC102, Pemetrexed Disodium, Cisplatin) - Phase I: Patients receive 50, 75 or 100 mg/day of TRC102 PO QD on days 1-4, 500 mg/m^2 of pemetrexed disodium IV over 10 minutes, and 60 or 75 mg/m^2 of cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue TRC102 and pemetrexed disodium beyond cycle 6 if the patient continues to benefit from treatment at the discretion of the treating physician.
- Arm B (TRC102, Pemetrexed Disodium) - Phase II: Patients receive 50 mg/day of TRC102 PO QD on days 1-4 and 500 mg/m^2 of pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue TRC102 and pemetrexed disodium beyond cycle 6 if the patient continues to benefit from treatment at the discretion of the treating physician.
Arm/Group | Arm A (TRC102, Pemetrexed Disodium, Cisplatin) - Phase I | Arm B (TRC102, Pemetrexed Disodium) - Phase II
Number analyzed (Participants) | 16 | 14
Months | 7.1 [1.4 to 14.4] | 3.8 [1.4 to 6.5]
Statistical Analysis 1: Comparison: Arm A (TRC102, Pemetrexed Disodium, Cisplatin) - Phase I vs Arm B (TRC102, Pemetrexed Disodium) - Phase II; Test type: Other; p = 0.08, Log Rank

5. Secondary Outcome: Overall Survival
Description: Overall survival will be summarized as time from first protocol treatment until death from any cause, using the product-limit Kaplan-Meier estimator.
Time Frame: From start of treatment to time of death from any cause, assessed up to at least 3 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (TRC102, Pemetrexed Disodium, Cisplatin) - Phase I | Arm B (TRC102, Pemetrexed Disodium) - Phase II
Number analyzed (Participants) | 16 | 14
Months | 20.0 [7.9 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 15.9 [3.4 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Arm A (TRC102, Pemetrexed Disodium, Cisplatin) - Phase I vs Arm B (TRC102, Pemetrexed Disodium) - Phase II; Test type: Other; p = 0.15, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of initial treatment until 30 days post discontinuation of treatment, up to 5 years.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Groups:
- Arm A, Dose Level 1 - 50mg TRC102, 60mg/m^2 Cisplatin (Phase I): TRC102 50 mg PO days 1-4; Pemetrex 500 mg/m^2 IV over 10 min day1; Cisplatin 60 mg/m^2 IV over 30-60 min day1
- Arm A, Dose Level 2 - 75mg TRC102, 60mg/m^2 Cisplatin (Phase I): TRC102 75 mg PO days 1-4; Pemetrex 500 mg/m^2 IV over 10 min day1; Cisplatin 60 mg/m^2 IV over 30-60 min day1
- Arm A, Dose Level 3 - 100mg TRC102, 60mg/m^2 Cisplatin (Phase I): TRC102 100 mg PO days 1-4; Pemetrex 500 mg/m^2 IV over 10 min day1; Cisplatin 60 mg/m^2 IV over 30-60 min day1
- Arm A, Dose Level 4 - 100mg TRC102, 75mg/m^2 Cisplatin (Phase I): TRC102 100 mg PO days 1-4; Pemetrex 500 mg/m^2 IV over 10 min day1; Cisplatin 75 mg/m^2 IV over 30-60 min day1
- Arm B, Dose Level 1 - 50mg TRC102 (Phase II): TRC102 50mg PO on days 1-4; Pemetrex 500mg/m^2 IV over 10 min day 1
Arm/Group | Arm A, Dose Level 1 - 50mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 2 - 75mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 3 - 100mg TRC102, 60mg/m^2 Cisplatin (Phase I) | Arm A, Dose Level 4 - 100mg TRC102, 75mg/m^2 Cisplatin (Phase I) | Arm B, Dose Level 1 - 50mg TRC102 (Phase II)
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/4 | 2/3 | 0/6 | 6/14
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/4 | 2/3 | 3/6 | 9/14
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 6/6 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A, Dose Level 1 - 50mg TRC102, 60mg/m^2 Cisplatin (Phase I) (N=3) | Arm A, Dose Level 2 - 75mg TRC102, 60mg/m^2 Cisplatin (Phase I) (N=4) | Arm A, Dose Level 3 - 100mg TRC102, 60mg/m^2 Cisplatin (Phase I) (N=3) | Arm A, Dose Level 4 - 100mg TRC102, 75mg/m^2 Cisplatin (Phase I) (N=6) | Arm B, Dose Level 1 - 50mg TRC102 (Phase II) (N=14)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus/Enterovirus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A, Dose Level 1 - 50mg TRC102, 60mg/m^2 Cisplatin (Phase I) (N=3) | Arm A, Dose Level 2 - 75mg TRC102, 60mg/m^2 Cisplatin (Phase I) (N=4) | Arm A, Dose Level 3 - 100mg TRC102, 60mg/m^2 Cisplatin (Phase I) (N=3) | Arm A, Dose Level 4 - 100mg TRC102, 75mg/m^2 Cisplatin (Phase I) (N=6) | Arm B, Dose Level 1 - 50mg TRC102 (Phase II) (N=14)
Anemia (Blood and lymphatic system disorders) | 2 (11) | 3 (19) | 3 (70) | 6 (52) | 10 (89)
LDH Increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
nose bleed (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (5) | 1 (3) | 2 (3) | 1 (4) | 2 (4)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (6) | 1 (1) | 2 (3) | 1 (1)
Ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Flashing lights (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Unequal Pupil Dilation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (14)
discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
drooping right eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
unequal pupil dilation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (5) | 1 (2) | 1 (3) | 1 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (4)
Constipation (Gastrointestinal disorders) | 2 (7) | 2 (7) | 2 (27) | 5 (22) | 4 (21)
Dark stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (7) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (10)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (20) | 1 (11) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (3)
Green Stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Helicobactor Pylori Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (6) | 3 (11) | 3 (49) | 4 (33) | 5 (22)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (5) | 2 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (7) | 1 (2) | 2 (9) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (7) | 1 (13) | 1 (1) | 3 (9)
Fatigue (General disorders) | 2 (9) | 4 (29) | 3 (45) | 3 (35) | 7 (20)
Fever (General disorders) | 0 (0) | 1 (6) | 1 (3) | 2 (2) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (6)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (31)
night sweats (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
rhinorrhea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (6) | 0 (0)
CrCl decrease (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (4)
decrease CrCl (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (15)
decrecease CrCl (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALT decrease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AST decrease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (18) | 1 (8) | 3 (11) | 3 (4)
Alkaline phosphatase increased (Investigations) | 2 (3) | 1 (5) | 1 (13) | 2 (5) | 2 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (20) | 2 (14) | 2 (12) | 6 (22)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (14) | 0 (0) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (19) | 1 (3) | 1 (2) | 2 (12)
Flashing lights -eye (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LDH increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (17)
LDH increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (8)
Lymphocyte count decreased (Investigations) | 1 (10) | 2 (18) | 1 (18) | 4 (24) | 10 (58)
Neutrophil count decreased (Investigations) | 3 (8) | 2 (13) | 3 (9) | 1 (1) | 5 (14)
Platelet count decreased (Investigations) | 3 (12) | 2 (13) | 2 (11) | 1 (2) | 1 (13)
Weight gain (Investigations) | 1 (1) | 0 (0) | 1 (10) | 0 (0) | 1 (7)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 2 (2)
White blood cell decreased (Investigations) | 3 (18) | 3 (17) | 3 (8) | 2 (12) | 8 (40)
blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
decrease AST (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
decrease ALT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0)
decrease AST (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
decrese ALT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
elevated LDH (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
elevated LDh (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
elevated troponin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
increase LDH (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
incresae LDH (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
runny nose (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9)
total protein decrease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
transferrin saturation decrease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (12)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (8) | 4 (27) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated LDH (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (10) | 3 (17) | 1 (4) | 3 (24)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (11) | 1 (3) | 3 (20) | 8 (75)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5) | 1 (3) | 2 (25) | 1 (11) | 6 (16)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (13) | 0 (0) | 2 (7) | 6 (20)
Increased LDH (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Iron decrease (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
LDH (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
LDH Elevated (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Low Iron (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
decrease total protein (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hyponatrmia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
increased LDH (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
low iron (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (14) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 1 (13)
R. distal hand numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right Hand Numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
increased shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
truncal instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
soft tissue growth on right upper latera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (4) | 2 (8) | 4 (12) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (6) | 2 (12)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 2 (4)
Memory impairment (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (10) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (3) | 1 (2) | 2 (6) | 1 (1)
Right Distal Hand numbness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
disorientation (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
slow walking/speech (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (7)
Confusion (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (25) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (5) | 2 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (8) | 1 (7)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (16) | 2 (7) | 1 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5) | 1 (17) | 1 (4) | 5 (15)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 2 (27) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (4) | 0 (0) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
rhinnorhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritic rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
cellulitiis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
cellulittis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
skin rash on scalp (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
sore on lower lip (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 1 (2)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypertension (Vascular disorders) | 2 (8) | 1 (8) | 3 (26) | 2 (2) | 3 (21)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 1 (3) | 1 (6) | 2 (4)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (9)
Sweats (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (9) | 0 (0)
superficial thrombophlebitis greater sap (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT02535312/Prot_SAP_000.pdf